CLINICAL TRIAL: NCT03125369
Title: Prospective Randomized Trial Comparing Single Loop Duodenojejunal Bypass With Sleeve Gastrectomy Versus Standard Roux-en-Y Gastric Bypass in Patients With Poorly Controlled Type 2 Diabetes Mellitus: From Clinical Outcomes to Hormonal Mechanism
Brief Title: Single Loop DJB Sleeve Gastrectomy for Poorly Controlled T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Enders K.W. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLDJBSG_DM
Record Dates: First submitted 2016-04-29; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus; Obesity; Bariatric Surgery Candidate; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duodenojejunal bypass (Experimental): patients receive sleeve gastrectomy plus duodeno-jejunal bypass
  Interventions: Procedure: Sleeve gastrectomy + duodeno-jejunal bypass
- Roux-en-Y gastric bypass (Active Comparator): patients receive roux-Y gastric bypass
  Interventions: Procedure: Roux-Y gastric bypass

INTERVENTIONS:
Procedure: Sleeve gastrectomy + duodeno-jejunal bypass
  Arms: Duodenojejunal bypass
Procedure: Roux-Y gastric bypass
  Arms: Roux-en-Y gastric bypass

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic progressive illness affecting a substantial percentage of the general population. While pharmacotherapy remains the mainstay of treatment, around 60% of patients cannot achieve the recommended goals for diabetic control. Weight control is a well-known essential component in normalizing blood glucose level in T2DM. The term metabolic surgery is recently introduced and it is now increasingly accepted as a valid option for obese T2DM patients with poor glycemic control despite optimal medical therapy. While laparoscopic roux-en-Y gastric bypass (RYGBP) is the gold-standard bariatric/metabolic procedure in many countries, it is not widely accepted in Asia. Recently, a novel bypass technique called single loop duodenojejunal bypass with sleeve gastrectomy (SLDJB-SG) has been developed trying to tackle most drawbacks of RYGBP. Realizing there is a knowledge gap in applying the new duodenojejunal bypass procedure to obese T2DM patients, we propose to investigate and compare the efficacy of glycemic control and functional outcomes of SLDJB-SG with conventional RYGBP.

DETAILED DESCRIPTION:
Aim of study:

To investigate and compare the safety profile, functional outcomes, efficacy in diabetic control and changes of hormonal profile of laparoscopic single loop duodenojejunal bypass plus sleeve gastrectomy (SLDJB-SG) versus the conventional standard roux-en-Y gastric bypass (RYGBP).

Hypothesis:

The efficacy of glycemic control and functional outcomes of SLDJB-SG is better than conventional RYGBP, and is a more suitable option for obese Chinese diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 to 65 years
* at least 2 years of T2DM
* a BMI between 28 to 42 kg/m2
* a HbA1c level above 7% despite multiple oral medications (> 2) at higher than or equal to half-maximal dose, or already using insulin injection for more than 6 months
* no active cardiovascular diseases, and
* a ASA grade II or below
* a fasting C-peptide < 0.6ug/L

Exclusion Criteria:

* significant anaesthetic risk ASA grade III or above
* history of diabetic ketoacidosis
* uncontrolled DM with HbA1c > 12%
* malignancy diagnosed within 5 years
* chronic renal failure requiring dialysis
* previous upper abdominal surgery affecting gastroduodenal configuration
* major psychiatric illness including major depression and substance abuse
* pregnancy or ongoing breast-feeding
* inmates

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
% of patient achieve HbA1c<6% | 1 year

SECONDARY OUTCOMES:
operation time | during operation
Total blood loss | during operation
  Total blood loss data from operation record
Perioperative complications | 30 days
mortality | 30 days
Postoperative hospital stay | during index operation
Excessive body weight loss (kg) | 6 months & 1 year
BMI change (kg/m^2) | 6 months & 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Enders KW Ng, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided